CLINICAL TRIAL: NCT00339729
Title: Johnston County ADHD Study: Environmental, Reproductive and Familial Risk Factors for Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Johnston County ADHD Study: Environmental, Reporductive, and Familial Risk Factors for Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997029; OH97-E-N029
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-05-24

CONDITIONS: Attention-Deficit Hyperactivity Disorder
Keywords: Children; Behavior; Epidemiology; Lead; Learning Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Behavior; Learning Disabilities

SUMMARY:
We propose a population-based case-control study among 7000 elementary school children in semi-rural Johnston County, NC. Teachers will complete a screening form on each child. Controls will be randomly selected. Mothers of potential cases and controls will be interviewed by telephone about their child's symptoms of ADHD and exposure history, their family history of ADHD, and their reproductive and exposure history. Children's shed baby teeth will be analyzed for lead. Mothers will complete brief parenting scales and the Child Behavior Checklist. School records will be collected. The study goals are to identify risk factors for ADHD including preterm delivery and childhood lead exposure.

DETAILED DESCRIPTION:
We propose a population-based case-control study among 7000 elementary school children in semi-rural Johnston County, NC. Teachers will complete a screening form on each child. Controls will be randomly selected. Mothers of potential cases and controls will be interviewed by telephone about their child's symptoms of ADHD and exposure history, their family history of ADHD, and their reproductive and exposure history. Children's shed baby teeth will be analyzed for lead. Mothers will complete brief parenting scales and the Child Behavior Checklist. School records will be collected. The study goals are to identify risk factors for ADHD including preterm delivery and childhood lead exposure.

ELIGIBILITY:
* INCLUSION CRITERIA:

During the first phase of the study, all children will be screened by the homeroom teacher, EXCEPT for those students in certain self-contained classrooms. Self-contained classrooms for students with an IQ less than 70 or autism will be omitted from the screening. In the second phase of the study, children designated as "LEP", or Low English Proficiency, will be excluded from the study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8000
Dates: Start 1997-05-07; Study Completion 2007-05-24

CONTACTS AND LOCATIONS:
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States